CLINICAL TRIAL: NCT01033162
Title: Using Technology to Enhance Cancer Communication and Improve Clinical Outcome: Effectiveness of the CHESS Ehealth Cancer Support Intervention in Population-Based Care Study
Brief Title: Effectiveness of the CHESS eHealth Cancer Support Intervention in Population-based Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-2008-0222; 5P50CA095817 (NIH); XP08323 (Other: University of Wisconsin Carbone Cancer Center); NCI-2013-01101 (Registry Identifier: NCI Trial ID); A534253 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*G (Other: UW Madison)
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2016-02

CONDITIONS: Primary Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): A group using a Basic ICCS provided by KPNW
- Intervention (Experimental): A group using an enhanced ICCS with KPNW web resources and the Comprehensive Health Enhancement Support System (CHESS.)
  Interventions: Behavioral: Enhanced ICCS with KPNW web resources and the Comprehensive Health Enhancement Support System (CHESS.)

INTERVENTIONS:
Behavioral: Enhanced ICCS with KPNW web resources and the Comprehensive Health Enhancement Support System (CHESS.) — Half of the participating women will be randomly assigned to use an informative but static website (Basic ICCS), and half will be offered a fully interactive CHESS (Enhanced ICCS + the Basic ICCS). Study outcome data will be gathered from patients, clinicians, and the healthcare system (i.e., from the electronic medical record: EMR) for at least 8 months after study entry. We propose that the Enhanced ICCS relative to the Basic ICCS, will:
  * Improve patients' sense of cancer information competence (perceived ability to obtain and use relevant information)
  * Reduce patients' negative affect and increase their emotional well being
  * Improve patients' sense of social support
  * Improve patients' health self-efficacy
  * Improve patients' ratings of experience with cancer specialty care services
  * Improve patients' health related quality of life (HRQL)
  * Improve clinicians' ratings of quality of patient contacts
  * Reduce healthcare utilization and costs (obtained via the EMR)
  Arms: Intervention

SUMMARY:
The study's aim is to provide information about the clinical and business cases for comprehensive interactive cancer communication systems (ICCS) in the context of real world use for cancer care.

This study will be conducted within the Kaiser Permanente Northwest (KPNW) healthcare system. Outcomes for this study include amount of ICCS use and women's ratings of cancer information competence, perceived social support, and emotional well being. Secondary outcomes will include healthcare utilization, cost-effectiveness, and clinician ratings of healthcare visits.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be within 2 months of their primary breast cancer diagnosis,
* All subjects must be at least 18 years of age

Exclusion Criteria:

* Illiterate
* Homeless

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2009-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Amount of ICCS use and women's ratings of cancer information competence, perceived social support, and emotional well being. Secondary outcomes will include healthcare utilization, cost-effectiveness, and clinician ratings of healthcare visits. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Baker, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Kaiser Permanente Northwest, Portland, Oregon, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/